CLINICAL TRIAL: NCT01096615
Title: Evaluation of the Effect of Probiotic Lactobacillus Paracasei Lp-33 for the Management of Rhinitis in People Sensitized to Allergens. A Double Blind Randomized Parallel Placebo Controlled Study. (GA2LEN STUDY) BIONATLANTA Project
Brief Title: Effect Of Probiotic Lactobacillus Paracasei Lp-33 For The Management Of Rhinitis In People Sensitized To Allergens
Acronym: BionAtlanta
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Medication Familiale (Industry)
Collaborators: Chr Hansen A/S (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 13609
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Rhinitis
Keywords: Allergic rhinitis-Probiotic Lactobacillus paracasei LP-33-
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tested product: Lactobacillus paracasei LP-33 (Active Comparator): Each patient will be randomly assigned to either tested product or comparative product (placebo) in accordance with a randomisation table
  Interventions: Dietary Supplement: Lactobacillus paracasei LP-33
- Comparative product : placebo (Placebo Comparator): Each patient will be randomly assigned to either tested product or comparative product (placebo) in accordance with a randomisation table .
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Description:
  - capsule size 3
  Composition of the product:
  * 45 mg of microcristalline cellulose,
  * 132 mg of maltodextrin,
  * 3 mg of magnesium stearate.
  Composition of the capsule:
  * 46 mg of hypromellose,
  * 1 mg of titanium dioxide.
  Packaging:
  Products are packaged in aluminium tubes of 30 capsules.
  Storage:
  The product should be stored in a fridge. Direction for use: subject should consume 1 capsule daily together with a meal, with a glass of water.
  The study products will be consumed daily for 7 weeks.
  Arms: Comparative product : placebo
Dietary Supplement: Lactobacillus paracasei LP-33 — Description:
  * minimum 2.0x109 CFU of Lactobacillus paracasei LP-33
  * capsule size 3 1 capsule daily together with a meal, with a glass of water.
  Arms: Tested product: Lactobacillus paracasei LP-33

SUMMARY:
The aim of the study is to show an improvement of quality of life on the 5th week of product consumption (probiotic Lactobacillus paracasei LP-33)(as assessed by RQLQ global score) in subjects with persistent allergic rhinitis currently treated with Loratadine or oral anti-histaminic treatment.

DETAILED DESCRIPTION:
Oral H1-antihistamines are first treatment recommended for allergic rhinitis (Bousquet et al, 2008) however they do not completely alleviate symptoms. This new study will therefore assess the effect of Lactobacillus paracasei LP-33 in the management of nasal and ocular symptoms, in addition to H1-antihistamines treatment. The main objective is to evaluate the effect of Lactobacillus paracasei LP-33 on quality of life. Additionally allergic rhinitis symptoms (nasal and eye symptoms) and immunological parameters will be evaluated, before and during the supplementation. Lactobacillus paracasei LP-33 is targeting the general population and improving quality of life of people sensitized to allergens. The study will be conducted in Europe on adult subjects with persistent allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects;
* Aged 18 to 60 years;
* People with nasal and ocular discomfort at least sensitized to grass pollen;
* Subject with PER allergy (persistent form) as defined by ARIA guidelines or with a recurrent history of seasonal allergic rhinitis documented by treatment intakes in his medical dossier.
* Previous positive skin prick test or presence of specific serum IgE antibodies class II or above against timothy grass in the last 5 years. If no data are available, a test for detection of timothy grass specific serum IgE antibodies (Phadia CAP System) will be performed at the pre-inclusion visit;
* With RQLQ score ≥ 2;
* Subjects agree to stop consumption of probiotics (food or dietary supplement containing probiotics) and vitamins and/or minerals during the study (D-10/D-7 to D49).

Female subjects with efficient contraception and asthmatic subjects (with a controlled disease and without oral corticosteroid) can be included in the study.

The baseline period prior to treatment with Lactobacillus paracasei LP-33 is 7 days. On recommendations of the consulted experts, Pr Bousquet and Pr Hamelmann, a wash-out period of 3 additional days is recommended before baseline for subject using intranasal corticosteroid before their inclusion. As a consequence, the baseline may be extended to 10 days for these subjects In case the subject consumed an anti-H1 (other than Loratadine) before his (her) inclusion, he (she) will have to switch to Loratadine to be included.

Exclusion Criteria:

* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial;

  * Presenting a psychological incapability or having a bad comprehension of the language (French or German according to the concerned country) to understand the information letter and then to sign the informed consent;
  * Refusing to sign the informed consent;
  * Adult under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;
  * Pregnant or breastfeeding women;
  * Use of medication which could interfere with the study in the investigator's opinion (antibiotics, etc…);
  * Subject who does not agree to stop his/her consumption of dietary supplements and foods containing probiotics and his/her supplementation of vitamins/minerals during the study (D-10/D-7 to D49).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The primary criterion is the RQLQ global score measured at the end of Week 0 and Week 5. | Week 0 and Week 5
  The RQLQ includes 28 questions (completed between 10-15 min). Subjects are asked to recall their experiences during the previous week and to respond to each question on a 7-point scale (0 = no impairment, 6 = severe impairment). The RQLQ score ranges from 0 to 6. This questionnaire will be filled in by volunteers on D0 and D35.
  The aim of the study is to show an improvement of quality of life on the 5th week of product consumption (as assessed by RQLQ global score) in subjects with persistent allergic rhinitis currently treated with Loratadine or oral anti-histaminic treatment.

SECONDARY OUTCOMES:
To show a decrease in allergic rhinitis symptoms on the 5th week of product consumption (as assessed by RQLQ and RTSS-5) | Week 0-Week 5
To show an increase in the time of 1st exacerbation of symptoms of rhinitis symptom with Lactobacillus paracasei LP-33 | Week 5- Week 7

CONTACTS AND LOCATIONS:
Overall Officials: Jean BOUSQUET, Pr, Study Chair
Locations (125):
- France (125):
  - Corinne SION, Aix-en-Provence
  - Alain FAUDIN, Alès
  - Philippe PIAT, Alès
  - Sylvie CHABROL-RIVIERE, Alès
  - Daniel FERET, Aubevoye
  - Florian KOMAC, Aubord
  - Alain GIACOMINO, Avoine
  - Jean DEFLAUX, Beaucaire
  - Sébastien CONVENT, Beauvoisin
  - Catherine BRUNET-CAZOT, Béziers
  - Emmanuel DEJOUX, Béziers
  - Gabriel VENTURINI, Béziers
  - Nicolas BRETON, Béziers
  - Robert COMBET, Béziers
  - Thierry STEFANAGGI, Béziers
  - Olivier BISCH, Bischeim
  - Sabine GRUTTER, Bischeim
  - Sophie ROSENBERG, Bischeim
  - Jacques RAMBAUD, Bompas
  - Chantal MARTIN, Bouillargues
  - Catherine AYRAL, Boujan-sur-Libron
  - Laurence DAGES, Bourg-Achard
  - Dominique EDET, Bretteville-l'Orgueilleuse
  - Didier CADINOT, Broglie
  - François LE HINGRAT, Calvisson
  - Bernadette CHAUFFAILLE, Castelnau-le-Lez
  - Georges BINET, Castelnaudary
  - Hervé VILAREM, Castelnaudary
  - Gladys HAVARD, Clarensac
  - Marc GARCIA, Clarensac
  - Michel AMOUYAL, Codognan
  - Nicole FERRIER, Codognan
  - Philippe GRUJARD, Colombelles
  - Philippe HEUZE, Cournonsec
  - Gregoire MARTOCQ, Cournonterrac
  - Bruno DAUBIN, Coursan
  - Jean-Baptiste DE LEMOS, Damville
  - Marcel RUETSCH, Dessenheim
  - Christian DAUGENET, Équeurdreville-Hainneville
  - Gérard DUGNY, Évreux
  - Thierry CANALI, Évreux
  - Frédéric RENOU, Fécamp
  - Pascal MABIRE, Fleury-sur-Orne
  - Alain LION, Gambsheim
  - Raymond WESTERFELD, Hangenbieten
  - Gérard TELLIER, Hautot-sur-Mer
  - Marc BUR, Herlisheim
  - Jean Pascal SASTOURNE, Ille-sur-Têt
  - Reinhard RENNER, Laroque-des-Albères
  - Christian FLAISSIER, Lasalle
  - Irène LAFONT, Lasalle
  - Patrick DUTILLEUL, Le Cailar
  - Claude BRUNAUD, Lignan-sur-Orb
  - Jean-Philippe RICHTER, Lingolsheim
  - Stéphane BOURGHOL, Marguerittes
  - Maurice GAY, Maurin
  - Patrick OLOMBEL, Mèze
  - Cécile BELIN-SAUGET, Montpellier
  - Jean François GUILLEM, Montpellier
  - Jean Roch ALEA, Montpellier
  - Marie Pascale DEMOLY, Montpellier
  - MONGIN, Montpellier
  - Thierry AUTARD, Montpellier
  - Victor BASTIDE, Montpellier
  - Michel CHASSAGNE, Montpellier
  - Philippe CAYRON, Montpellier
  - Jean Pierre CANO, Montpellier
  - Patrick VOGT, Mulhouse
  - Jean-Louis WURTZ, Mundolsheim
  - Nasser GOUCHENE, Nîmes
  - Paul REGNIER-VIGOUROUX, Nîmes
  - Claude BERNAT, Nîmes
  - Dominique BLOT, Nîmes
  - Marie Christine BONS-GALLET, Nîmes
  - Philippe IMBERT, Nîmes
  - COSTA, Nîmes
  - Georgios MARKIDIS, Obernai
  - Natacha HEITZ, Obernai
  - Yves-Olivier SCHLECHT, Obernai
  - Guy BIRRY, Ottrott
  - Bernard PRIJAC, Pacy-sur-Eure
  - Alain GUERRI, Perpignan
  - Chantal MALZAC, Perpignan
  - Gérard BOURREL, Perpignan
  - Serge ELIE, Pompignan
  - Sonia COURTOIS, Pont-de-l'Arche
  - Bernard GABBAI, Pont-Saint-Esprit
  - Geneviève DURANT, Rivesaltes
  - Baudoin PINSON, Rouen
  - Olivier BAISSAS, Rouen
  - Dominique GENOUD, Rousson
  - Sylvie OLLIVIER, Rousson
  - Patrick VERDAVOINE, Rugles
  - Béatrice LOGNOS-FOLCO, Saint-Georges-dOrques
  - Catherine MERCEY, Saint-Génis-des-Fontaines
  - Yves MERCEY, Saint-Génis-des-Fontaines
  - Jean-Yves DOERR, Saint-Sébastien-de-Morsent
  - Martine FERRE, Saint-Siffret
  - Gil MEYRAND, Sainte-Anastasie
  - Jean Baptiste THIBERT, Salses-le-Château
  - Léa ABOAF, Schilttigheim
  - Monique LESCOUTE, Schilttigheim
  - Raymond ATTUIL, Schilttigheim
  - Luc ECHINARD, Sète
  - Laurent TENNEZE, Sommières
  - Charles LOUSQUI, Strasbourg
  - Claire PFRUNNER-SCHNEIDER, Strasbourg
  - Claire ROLLAND-JACQUEMIN, Strasbourg
  - Hélène STURCHLER, Strasbourg
  - Joël ETIENNEZ, Strasbourg
  - Judah TOLEDANO, Strasbourg
  - Nathan ABENHAIM, Strasbourg
  - Patrick KORMANN, Strasbourg
  - Philippe MARMOR, Strasbourg
  - Roland BENEDIC, Strasbourg
  - Véronique PEREZ, Strasbourg
  - Maxime BOUMANDIL, Strasbourg
  - Hervé MOREL, Tilly-sur-Seulles
  - Bernard CLARY, Trèbes
  - Jacques GRAVES, Trèbes
  - Christian GIRARD, Uchaud
  - Eric LIOTARD, Uchaud
  - Olivier CHAIX, Uzès
  - François BAYLE, Valleraugue
  - Philippe BOISSON, Villé